CLINICAL TRIAL: NCT06353724
Title: Comparison Between the Effect of Using Conventional and Digital Oral Positional Radiation Stent on Healthy Tissues, Salivary PH
Brief Title: Comparison Between the Effect of Using Conventional and Digital Oral Positional Radiation Stent
Acronym: stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Samar Hesham Maklad, Teaching assistant at faculty of dentistry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RP2218
Record Dates: First submitted 2024-03-20; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Radiotherapy Side Effect
Keywords: Radiation; Positioning stent; Removable prosthesis
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional positioning stent (Placebo Comparator): The Oral positioning stent were constructed according to the conventional technique
  Interventions: Device: conventional oral positioning stent were used during radiation planning and the PTV will be defined and contoured in computed tomography pre irradiation planning
- Digital positioning stent (Active Comparator): The Oral positioning stent will be constructed digitally
  Interventions: Device: Digital positioning stent

INTERVENTIONS:
Device: conventional oral positioning stent were used during radiation planning and the PTV will be defined and contoured in computed tomography pre irradiation planning — Dosimetric analysis: the maxilla (area of the teeth), both parotid glands (ipsilateral and contralateral), the mandible, and the PTV were defined and contoured in computed tomography pre irradiation planning. The mean corresponding dose of each structure were acquired using a dose-volume histogram.
  All patients will complete the radiotherapy sessions using the positional radiation prosthesis.
  Mucositis assessment: The severity of mucositis will be assessed weekly from the beginning of RT to the end of the treatment (mean time, 7 weeks). It will be scored in accordance with the classification criteria of the National Cancer Institute.
  PH of saliva measurement: Collection of saliva sample were done from each patient to measure salivary PH by digital PH meter before beginning of radiotherapy and the measurement will be continued weekly till the end of the treatment.
  Arms: conventional positioning stent
Device: Digital positioning stent — Digital positioning stent
  Arms: Digital positioning stent

SUMMARY:
The goal of this clinical trial is to compare between the Effect of Using Conventional and Digital Oral Positional Radiation Stent on Healthy tissues, salivary PH. The main question it aims to answer are: Does the difference in manufacturing method affect on Healthy tissues, salivary PH.

Participants will use radiation positioning stent during radiotherapy sessions Two groups will be compared

* Group A: OPRS was constructed according to the conventional technique.
* Group B: OPRS was constructed digitally using CAD /CAM technology. to evaluate Dosimetric analysis to quantify the radiation dose in OARs, PH of saliva measurement and Mucositis assessment.

DETAILED DESCRIPTION:
This study will be a clinically prospective study that will include 16 patients with head and neck cancer. This study will be carried out at the Clinical Prosthodontics Department & Clinical Oncology Department of Tanta University.

Informed consent will be obtained from all patients with maintenance of their privacy prior to inclusion in the study according to the guidelines on human research adopted by the Research Ethics Committee, Faculty of Dentistry, Tanta University.

Patient's evaluation:

All patients will be subjected to the following protocol:

Oral examination: Clinical dental evaluation, intraoral photography and mouth opening measurements

Grouping: The patients will be divided randomly into 2 groups (each group consists of 8 patients) according to the technique that will be used for construction:

First group: The OPRS will be constructed according to the conventional technique.27

Second group: The OPRS will be constructed digitally according to the following steps:

Intraoral scanning: It will be done using an intraoral scanner to generate three 3D images: the first of the superior arch, the second of the inferior arch, and the third of the maximum habitual intercuspation. Images will be compiled into a 3D file system.

Oral positioning radiation stent design: The compiled file will be exported into Exocad software, which is smart software for dental design on digital models, for stent design, and by using a virtual articulator.

3D printing: After optimizing the digital file, 3D printing will be performed. The oral positioning radiation stent will be printed using the 3D printer Resin Printing Material.

For both groups:

Insertion: making the necessary adjustment will be done.

RT techniques and dose distributions:

All patients will be referred to the RT department for IMRT planning. During the pre-irradiation simulation, the intraoral stents will be placed, and the patients will be immobilized by individual thermoplastic masks. A computed tomography scan will be conducted to determine the precise planning target volume (PTV); all patients will be scanned using the positional prosthesis once and without it.

Dosimetric analysis:

To quantify the radiation dose in the structures, the maxilla (area of the teeth), both parotid glands (ipsilateral and contralateral), the mandible, and the PTV will be defined and contoured in computed tomography pre-irradiation planning. The mean corresponding dose of each structure will be acquired using a dose-volume histogram.

All patients will complete the radiotherapy sessions using the positional radiation prosthesis together with the extra oral immobilization masks.

Mucositis assessment:

The severity of mucositis will be assessed weekly from the beginning of RT to the end of the treatment (mean time, 7 weeks). It will be scored in accordance with the classification criteria of the National Cancer Institute.

PH of saliva measurement:

A saliva sample will be collected from each patient to measure salivary PH by digital PH meter 19 before the beginning of radiotherapy, and the measurement will be continued weekly until the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Limit of age was between 20 -40 years old.
* Inter-arch distance ≥ 1.5 cm
* Good oral hygiene.

Exclusion Criteria:

* Patients with conditions that limited the construction of the stent (e.g. gross tumor block most of the oral cavity, sever limited mouth opening)
* Patients with recurrent cancerous lesions.
* Edentulous patients.
* Previously radiotherapy for head and neck
* Smoking.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Dosimetric analysis | 1 week
  The teeth away from the target site, both parotid glands and the maxilla, and OARs were defined and contoured in CT pre-irradiation planning using ECLIPSE software to each patient with the stent and without it and the mean corresponding dose of each structure was acquired using a dose volume histogram (DVH).
PH of saliva measurement: | 4 weeks
  Salivary PH was measured by digital PH meter before beginning of RT and the measurement was continued weekly throughout the treatment period till its end.
Mucositis assessment: | 4 weeks
  The severity of mucositis was assessed weekly from the beginning of RT to the end of the treatment at the RT department. The grading was scored in accordance with the Mucositis grading of National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), grading scores from 0-4 which 0 means better (None) and 4 means worse (Necrosis or deep ulceration; may include bleeding not induced by minor trauma or abrasion)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No